CLINICAL TRIAL: NCT00759278
Title: A Comparison of Fetal Hemodynamic Measurements Between Pregnant Women Taking Anti-hypertensive Medication and Controls
Brief Title: Comparison Fetal Hemodynamic Measurements Antihypertensive Versus Control
Status: Withdrawn | Type: Observational
Why Stopped: No participants
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, FolkJ, Associate Professor, State University of New York - Upstate Medical University
Other Study IDs: IRBPHS 5215
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Hypertension; Pregnancy
Keywords: pregnancy; umbilical artery systolic to diastolic flow ratio; middle cerebral artery peak systolic flow; antihypertensive medication
MeSH Terms: conditions — Hypertension | interventions — Pregnancy; High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Group of 30 women who are pregnant as subjects that take antihypertensive medication
  Interventions: Procedure: ultrasound evaluation in pregnancy
- 2: Group of 30 women who are pregnant and do not take antihypertensive medications as a control group
  Interventions: Procedure: ultrasound evaluation in pregnancy

INTERVENTIONS:
Procedure: ultrasound evaluation in pregnancy — Subjects enrolled will have a series of ultrasound evaluations to assess parameters in the study. Ultrasound is a non-invasive technique for creating images that does not use radiation and is routine in obstetrical practice
  Other Names: Sonogram

SUMMARY:
This is a prospective case-control study to evaluate women who are pregnant and take antihypertensive medication for fetal hemodynamics (middle cerebral artery peak systolic flow and umbilical artery Doppler systolic to diastolic ratio) compared to a control group of pregnant women not taking these kinds of medications. The hypothesis is that the investigators expect to observe little to no difference in the comparison between the medication group and the control group.

DETAILED DESCRIPTION:
Chronic hypertension is a common medical condition during pregnancy, occurring in up to 5 percent of pregnant women. There are significant maternal, fetal, and neonatal morbidity and mortality associated with this disease [1,2]. Chronic hypertension in pregnancy has been defined as elevated blood pressure detected and confirmed before the 20th week of gestation or hypertension present prior to conception. Chronic hypertension is usually classified as mild with systolic blood pressure greater than or equal to 140 mmHg or diastolic blood pressure greater than or equal to 90 mmHg. Severe hypertension is defined as systolic blood pressure greater than or equal to 180 mmHg or diastolic blood pressure greater than or equal to 110 mmHg [3]. Adverse outcomes associated with chronic hypertension in pregnancy include preterm delivery, intrauterine growth restriction (IUGR), intrauterine fetal demise (IUFD), placental abruption, and cesarean delivery [4]. The incidence of superimposed preeclampsia has been reported in up to 50 percent of women with severe chronic hypertension [5]. Many of these women have medical management with anti-hypertensive medications during pregnancy. Data is lacking regarding improvement in neonatal outcome, and there is evidence that anti-hypertensive medications may interfere with uteroplacental blood flow and fetal growth [3,6]. Despite a lack of support in the literature for medication in the management of hypertension in pregnancy, current recommendations recognize a role for medication use for at least severe chronic hypertension [1].

The umbilical arteries arise within fetal circulation from the common iliac arteries and represent the dominant circulatory outflow of the distal aortic circulation and contribute entirely to placental circulation. Normal umbilical artery resistance to blood flow progressively decreases throughout pregnancy, reflecting the progressive increase in placental mass and the increased numbers of tertiary villous small vessels of the placenta [7]. Doppler ultrasonography is a noninvasive technique that is used to assess the hemodynamic components of vascular impedance within the placenta. Umbilical artery Doppler flow velocimetry has been developed to evaluate fetal condition en-utero [8]. Normally developing and growing fetuses are characterized by high velocity diastolic umbilical artery flow, while those with IUGR have decreased, absent, or reversed diastolic flow [9,10]. Abnormal umbilical artery flow has been defined as the presence of absent or reversed end diastolic flow or a flow index greater than two standard deviations above the reported mean flow index for a given gestational age [11,12]. Evaluation of umbilical artery hemodynamics is indicated as part of standard care when IUGR or significant fetal anemia due to iso-immunization is suspected [7,8].

A group of patients with pregnancies complicated by pregnancy-induced hypertension (PIH) were treated with anti-hypertensive drugs labetalol and nifedipine. These subjects had umbilical artery Doppler flow velocity and resistance index measurements at 27-32 weeks gestation and again at 33-36 weeks gestation. An increase in resistance index measurements was noted over time. The authors attributed this increase in umbilical artery resistance to progression in placental impairment due disease progression rather than the medication management of PIH [13]. Another group of patients with pregnancies complicated by preeclampsia had significantly elevated umbilical artery systolic flow to diastolic flow (S/D) ratios compared to a control group. When treated with an antihypertensive agent alpha-methyldopa, there was a significant reduction in umbilical artery S/D ratios in the group of women with preeclampsia [14]. An in-vitro study was undertaken with isolated segments of human umbilical cords that were evaluated for measured umbilical artery resistance. The segments were exposed to varying concentrations of common substances that affect arterial tone and are used as antihypertensive agents such as labetalol, alpha-methyldopa, nifedipine, and magnesium sulfate. All except alpha-methyldopa demonstrated a dose-dependant reduction in umbilical artery resistance due to direct umbilical artery smooth muscle relaxation [15].

The purpose of this study is to obtain information regarding umbilical and middle cerebral artery hemodynamics during pregnancies complicated by chronic hypertension managed with anti-hypertensive medication and compare the measured values obtained to pregnancies not complicated by chronic hypertension. We postulate that the use of anti-hypertensive agents during pregnancy do not significantly affect umbilical artery Doppler flow and middle cerebral artery peak systolic velocity measurements.

Specific Objectives:

1. Establish a cohort of subjects that have a history of chronic hypertension requiring anti-hypertensive medication during pregnancy to act as a study group
2. Establish a cohort of subjects that do not have chronic hypertension and do not take anti-hypertensive medication during pregnancy to act as a control group
3. Obtain standard measurements of utero-placental function on two occasions during the third trimester of pregnancy, the first between 26 to 33 weeks gestation and the second between 34 and 40 weeks gestation
4. The measurements of utero-placental function to include estimated fetal weight, average gestational size, amniotic fluid index, umbilical artery S/D ratio, and middle cerebral arterial peak velocity
5. Compare the results of measurements made in both groups at two different times in the third trimester of pregnancy to define differences potentially attributable to medication use during pregnancy
6. Use the results of this preliminary study to estimate how many subjects would be required to identify a statistically significant difference in fetal hemodynamic measurements potentially attributable to anti-hypertension agent use

Study Design:

This study will employ a prospective case-control design. A group of women with a history of chronic hypertension managed with anti-hypertensive medication will be identified as potential subjects for the study cohort. Each potential subject will have an assessment of her hypertension history, management, and associated vascular complications. A detailed review of her complete medical, surgical, gynecologic, and obstetrical history will be obtained as dictated by standard care. Appropriate management for each potential subject's medical and obstetrical condition will be provided according to accepted practice. Potential subjects for this cohort will be obstetrical patients cared for at the Regional Perinatal Center, Division of Maternal Fetal Medicine, Department of Obstetrics & Gynecology, SUNY Upstate Medical University.

A second group of women with no history of chronic hypertension will be identified as potential subjects for the control cohort. Each potential subject will have a detailed review of her complete medical, surgical, gynecologic, and obstetrical history will be obtained as dictated by standard care. Appropriate management for each potential subject's medical and obstetrical condition will be provided according to accepted practice. Potential subjects for this cohort will be obstetrical patients cared for at the Regional Perinatal Center, Division of Maternal Fetal Medicine, Department of Obstetrics & Gynecology, SUNY Upstate Medical University.

The subjects enrolled in both cohorts are seen at the Regional Perinatal Center for management of high-risk pregnancies. As part of intensified obstetrical care, ultrasound evaluation of interval fetal growth with an assessment of estimated fetal weight, average gestational size, and amniotic fluid index is standard around 28 weeks gestation and again at about 35 weeks gestation. Umbilical artery Doppler studies are usually reserved for fetuses with a diagnosis of suspected intrauterine growth restriction. Fetal middle cerebral artery peak flow velocity studies are usually reserved for suspected severe fetal anemia and have been used on an investigational basis for suspected intrauterine growth restriction. We anticipate most subjects will not have a pregnancy complicated by IUGR, therefore performing Doppler studies for umbilical artery S/D ratio and middle cerebral arterial peak velocity will not be standard care. Data will be collected in a database in a single computer on site at the Regional Perinatal Center. This computer is password protected and reserved for use by care providers at the Perinatal Center that will be investigators for this study. The database will record specific patient identifiers including subject name and chart number. These specific identifiers will be removed at the completion of data collection prior to data analysis.

Statistical Methods, Data Analysis, Interpretation:

There are few studies published regarding the use of anti-hypertensive agents during pregnancy and the effect of these agents on umbilical artery hemodynamics. These few studies usually involved 20 to 30 subjects. At this point, there is not enough information to estimate how many subjects would be required to measure a statistically significant difference potentially attributable to the use of these agents. For this preliminary study, we will obtain 30 subjects for the study cohort and 30 subjects for the control cohort. It is anticipated that it will take approximately one year to complete this study.

Once data collection is complete as described above, a comparison of means will be undertaken for umbilical artery Doppler studies between the two cohorts at the first and then again for the second gestational age measurements.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. A diagnosis of chronic hypertension by at least one of these criteria including hypertension that has persisted beyond the postpartum time frame of a prior pregnancy, hypertension diagnosed and managed before current pregnancy, or elevated blood pressure (systolic blood pressure > or = 140 mmHg or diastolic blood pressure > or = 90 mmHg) prior to 20 weeks gestation requiring medication management
3. Taking medication for control of chronic hypertension prior to study entry
4. Potential subjects taking medications for control of cardiac arrythmia that fall into the anti-hypertensive class will be considered for this cohort

Potential subjects for the control cohort:

1. At least 18 years of age
2. Absence of a diagnosis of chronic hypertension
3. Not taking medication for control of chronic hypertension or arrythmia

Exclusion Criteria:

1. Less than 18 years of age
2. Pregnancy complicated by significant fetal chromosomal anomaly, severe or multiple fetal anomalies, early onset amniotic fluid abnormalities, preterm labor, placental abruption, or IUGR
3. Inability to complete the informed consent process or participate in the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with established singleton pregnancy at least 18 years of age, with diagnosis of chronic hypertension or with no diagnosis of hypertension
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Fetal ultrasound assessment of middle cerebral artery and umbilical artery blood flow | 26 to 33 weeks gestation and 34 to 40 weeks gestational age

CONTACTS AND LOCATIONS:
Overall Officials: John J Folk, M.D., Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- Regional Perinatal Center University Health Care Center, Syracuse, New York, United States

REFERENCES:
- [Background] Gilstrap LC, Ranin SM. Chronic hypertension in pregnancy. ACOG Practice Bulletin July 2001; 29.
- [Background] Haddad B, Sibai BM. Chronic hypertension in pregnancy. Ann Med. 1999 Aug;31(4):246-52. doi: 10.3109/07853899908995887. PMID 10480755
- [Background] National High Blood Pressure Education Program Working Group Report on High Blood Pressure in Pregnancy. Am J Obstet Gynecol. 1990 Nov;163(5 Pt 1):1691-712. doi: 10.1016/0002-9378(90)90653-o. PMID 2104525
- [Background] Ferrer RL, Sibai BM, Mulrow CD, Chiquette E, Stevens KR, Cornell J. Management of mild chronic hypertension during pregnancy: a review. Obstet Gynecol. 2000 Nov;96(5 Pt 2):849-60. doi: 10.1016/s0029-7844(00)00938-8. PMID 11094241
- [Background] Sibai BM, Anderson GD. Pregnancy outcome of intensive therapy in severe hypertension in first trimester. Obstet Gynecol. 1986 Apr;67(4):517-22. PMID 3960423
- [Background] von Dadelszen P, Ornstein MP, Bull SB, Logan AG, Koren G, Magee LA. Fall in mean arterial pressure and fetal growth restriction in pregnancy hypertension: a meta-analysis. Lancet. 2000 Jan 8;355(9198):87-92. doi: 10.1016/s0140-6736(98)08049-0. PMID 10675164
- [Background] Harman CR. Chapter 21 Assessment of fetal health. Creasy RK, Resnik R, Iams JD (eds)Maternal-Fetal Medicine: Principles and Practice, 5th Edition. 2004; Saunders, Philadephia, Pennsylvania, 372.
- [Background] Rouse DJ. Antepartum fetal surveillance. ACOG Practice Bulletin, October 1999; 9.
- [Background] Erskine RL, Ritchie JW. Umbilical artery blood flow characteristics in normal and growth-retarded fetuses. Br J Obstet Gynaecol. 1985 Jun;92(6):605-10. doi: 10.1111/j.1471-0528.1985.tb01399.x. PMID 4005201
- [Background] Reuwer PJ, Bruinse HW, Stoutenbeek P, Haspels AA. Doppler assessment of the fetoplacental circulation in normal and growth-retarded fetuses. Eur J Obstet Gynecol Reprod Biol. 1984 Nov;18(4):199-205. doi: 10.1016/0028-2243(84)90117-5. PMID 6240422
- [Background] Trudinger BJ, Cook CM, Giles WB, Connelly A, Thompson RS. Umbilical artery flow velocity waveforms in high-risk pregnancy. Randomised controlled trial. Lancet. 1987 Jan 24;1(8526):188-90. doi: 10.1016/s0140-6736(87)90003-1. PMID 2880017
- [Background] Omtzigt AM, Reuwer PJ, Bruinse HW. A randomized controlled trial on the clinical value of umbilical Doppler velocimetry in antenatal care. Am J Obstet Gynecol. 1994 Feb;170(2):625-34. doi: 10.1016/s0002-9378(94)70240-3. PMID 8116724
- [Background] Gazzolo D, Visser GH, Russo A, Scopesi F, Santi F, Bruschettini PL. Pregnancy-induced hypertension, antihypertensive drugs and the development of fetal behavioural states. Early Hum Dev. 1998 Jan 9;50(2):149-57. doi: 10.1016/s0378-3732(97)00033-7. PMID 9483388
- [Background] Gunenc O, Cicek N, Gorkemli H, Celik C, Acar A, Akyurek C. The effect of methyldopa treatment on uterine, umblical and fetal middle cerebral artery blood flows in preeclamptic patients. Arch Gynecol Obstet. 2002 Jul;266(3):141-4. doi: 10.1007/s004040100214. PMID 12197552
- [Background] Houlihan DD, Dennedy MC, Ravikumar N, Morrison JJ. Anti-hypertensive therapy and the feto-placental circulation: effects on umbilical artery resistance. J Perinat Med. 2004;32(4):315-9. doi: 10.1515/JPM.2004.058. PMID 15346815